CLINICAL TRIAL: NCT01891058
Title: A Randomized, Controlled Comparison of Electrical Versus Pharmacological Cardioversion for Emergency Department Patients With Recent-Onset Atrial Fibrillation and Flutter (RAFF)
Brief Title: Trial of Electrical Versus Pharmacological Cardioversion for RAFF in the ED
Acronym: RAFF-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 20130331; G-13-0002756 (Other: Heart and Stroke Foundation)
Record Dates: First submitted 2013-06-19; First posted 2013-07-02 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drug-shock vs shock only (Active Comparator): For ED patients with RAFF, Investigators will compare conversion to normal sinus rhythm between the two strategies of i) attempted pharmacological cardioversion with intravenous procainamide followed by DC cardioversion if necessary (Drug-Shock), and ii) DC cardioversion alone (Shock Only).
  Interventions: Device: drug-shock vs shock only
- pad positions (No Intervention): For ED RAFF patients undergoing DC cardioversion, Investigators will compare conversion to normal sinus rhythm between the i) antero-posterior and ii) antero-lateral pad positions.

INTERVENTIONS:
Device: drug-shock vs shock only — procainamide followed by electrocardioversion if necessary vs cardioversion only.
  Arms: drug-shock vs shock only

SUMMARY:
Atrial fibrillation (AF) and atrial flutter (AFL) are cardiac rhythm problems where there is an irregular, rapid heart rate. Investigators plan to study Emergency Department (ED) patients with recent-onset episodes of AF or AFL (RAFF) where rapid heart rate requires urgent treatment to restore normal heart rhythm. RAFF is the most common rhythm disorder managed in the ED. Investigators recently showed that doctors use a wide variety of treatment approaches in Canadian EDs for RAFF. Also, the Canadian Cardiovascular Society Guidelines indicate that there have not been enough studies to know if the best treatment is to use an electrical shock (Shock Only) or drugs followed by shock (Drug-Shock). Investigators believe that Drug-Shock approach will be more effective and will help avoid an electric shock for many patients. Investigators also do not know if electrical shocks should be given with the electrode pads on the front (antero-lateral) or front and back (antero-posterior).

Investigators intend to conduct 2 randomized protocols within one study (partial factorial design) in order to answer these two questions. 1. Will initial drug treatment followed by electrical shock if necessary (Drug-Shock) lead to more patients being converted to normal heart rhythm than a strategy of only electrical shock (Shock Only)? 2. Will the antero-posterior pad position be more effective than the antero-lateral position? Investigators plan to enroll 468 RAFF patients at 8 large Canadian EDs. Patients will be randomized to 1 of 2 arms for each of the two protocols. Investigators primary outcome will be conversion to normal heart rhythm. Other outcomes will include heart rhythm at discharge, need for hospital admission, length of stay in ED, adverse events, patient satisfaction, and 14-day follow-up status.

Investigator results will add important information about the best and safest ways to treat RAFF patients in Canadian EDs. Ultimately Investigators expect to see fewer patients admitted to hospital and more patients rapidly and safely returned to their normal activities.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is characterized by disorganized atrial electrical depolarization leading to an irregular and rapid heart rate and is the most common arrhythmia seen in the emergency department (ED). Atrial flutter (AFL) is a less common arrhythmia with similar pathophysiology. Investigators will focus on recent-onset episodes of AF and AFL (RAFF), which have usually been present less than 48 hours, are highly symptomatic, and may be a first or recurrent event. There is a surprising lack of evidence regarding many important ED RAFF management questions and the 2011 Canadian Cardiovascular Society AF Guidelines indicate clinical equipoise for most facets of early care. In Canadian EDs, most physicians use the rhythm control approach, where attempts are made to cardiovert patients to sinus rhythm in the ED, either pharmacologically or electrically (DC cardioversion). Canadian ED physicians seem equally divided between those who prefer to attempt rhythm control initially with drugs and then move to DC cardioversion if necessary (Drug-Shock strategy) and those who prefer to start immediately with DC cardioversion (Shock Only strategy). Investigators recently completed a prospective cohort RAFF study (N=1,065, funded by the Heart and Stroke Foundation of Ontario) at 6 Canadian EDs. 73.3% of all patients underwent ED rhythm control with 34.4% receiving rhythm control drugs first and 38.9% receiving electrical shock first. There is also much variation in whether the DC cardioversion electrodes are placed in the front and back (antero-posterior) or front and side (antero-lateral) position (Figure 1).

Investigators believe that the Drug-Shock strategy has many advantages over a Shock Only strategy. Most Canadian EDs have a single physician on duty, which is a barrier to safe procedural sedation and DC cardioversion. Even in larger EDs, DC cardioversion requires 4 professional staff, has a risk associated with sedation, and can be frightening for patients. Investigators expect that the Drug-Shock strategy will be more effective because procainamide will facilitate DC cardioversion and prevent early return of AF. Even if the Drug-Shock strategy is not more effective overall, its use can prevent the need for DC cardioversion in 50-60% of patients. Regarding DC cardioversion pad placement, no randomized trials have ever been done with RAFF patients using modern biphasic devices at high energy levels.

Study Objectives: Investigators primary aim is to compare conversion to sinus rhythm between the strategies of i) attempted pharmacological cardioversion with intravenous procainamide followed by DC cardioversion if necessary (Drug-Shock) and ii) DC cardioversion alone (Shock Only). Investigators secondary aim is to compare the effectiveness of the i) antero-posterior and ii) antero-lateral pad positions.

Methods: Design and Interventions: Investigators propose a partial factorial study design with 2 protocols (Figure 2). All patients will participate in Protocol 1 (N=468) and most in Protocol 2 (N=356). 1. Drug versus Shock Protocol. This will be a randomized, blinded, placebo-controlled comparison of: i) attempted pharmacological cardioversion with intravenous procainamide (15mg/kg over 30 minutes) followed by DC cardioversion (200 joules x 3) if necessary (Drug-Shock), and ii) only DC cardioversion (Shock Only) (Hypothesis 1). 2. Pad Position Protocol. For the subset of patients who undergo DC cardioversion, this will be a randomized, open-label comparison of i) the antero-posterior pad position, and ii) the antero-lateral pad position (Hypothesis 2). Management protocols will be standardized. Randomization will be stratified by site and by rhythm (AF or AFL). Setting: 8 EDs of large, tertiary care Canadian hospitals. Subjects: Stable patients with primary diagnosis of RAFF where acute rhythm control is a safe option. Investigators will obtain patient consent. Outcomes: The primary outcome measure will be conversion to sinus rhythm and maintenance of sinus rhythm for at least 60 minutes; other outcomes will include sinus rhythm at discharge, hospital admission, length of stay in ED, adverse events, patient satisfaction, and 14-day follow-up status. Patients will be telephoned at 6 months and 1 year after the original ED visit to determine stroke-free status and medication changes. Data Analysis: Primary analysis will be intention-to-treat using chi-square testing. Sample Size: Investigators will require 213 evaluable patients per group to detect a minimal clinically important absolute difference of 10% between groups. Allowing for 10% non-compliance, investigators plan to enroll 468 patients.

Importance: This study will answer two important questions about the early management of ED RAFF patients, leading to higher rhythm conversion rates and lower admission rates. The results will inform future efforts to create effective, safe, and efficient pathways for RAFF patient management in Canada.

ELIGIBILITY:
Inclusion Criteria:

* include stable (see below) patients presenting with an episode of RAFF of at least 3 hours duration,
* where symptoms require urgent management and where pharmacological or DC cardioversion is a reasonable option because there is a clear history of:
* onset within 48 hours, or
* onset within 7 days and adequately anticoagulated for > 4 weeks (warfarin and INR > 2.0 or newer oral anticoagulants [dabigatran, rivaroxaban, and apixaban]), or
* onset within 7 days and no left atrial thrombus on TEE. Of note, Investigators will not exclude patients with prior episodes of RAFF.

Exclusion Criteria:

Investigators will exclude patients for the reasons listed below.

* who are unable to give consent;
* who have permanent (chronic) AF;
* whose episode did not clearly start within 48 hours [or 7 days if anticoagulated / normal TEE];
* who are deemed unstable and require immediate cardioversion: i) systolic blood pressure <100 mmHg; ii) rapid ventricular preexcitation (Wolff-Parkinson-White syndrome); iii) acute coronary syndrome - chest pain and acute ischemic changes on ECG; or iv) pulmonary edema - severe dyspnea requiring immediate IV diuretic, nitrates, or BIPAP;
* whose primary presentation was for another condition; examples include pneumonia, pulmonary embolism, and sepsis;
* who convert spontaneously to sinus rhythm prior to randomization; or
* who were previously enrolled in the study.

Safety Exclusions:

1. who are known to have severe heart failure (left ventricular ejection fraction <30% or have clinical or radiological evidence of acute HF);
2. whose heart rate < 55 bpm;
3. who have 3rd degree AV block or complete LBBB or a history of 2nd or 3rd degree AV block (in the absence of a permanent pacemaker or implantable cardioverter-defibrillator [ICD]);
4. whose ECG shows QTc >460ms;
5. who have Brugada syndrome (genetic disease with increased risk of sudden cardiac death);
6. who currently take class I or III antiarrhythmic drugs (last dose < 5 half-lives before enrolment) except Amiodarone;
7. who have hypersensitivity to procainamide, procaine, other ester-type local anesthetics, or any component of the formulation;
8. who have had a recent myocardial infarction (< 3 months);
9. who have these chronic diseases: renal failure (GFR <60 mL/min/1.73m2) or liver disease; or
10. who are breast feeding or pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2013-07-18 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
conversion to sinus rhythm | one year
  The primary outcome for both hypotheses will be conversion to sinus rhythm following randomization and maintenance of sinus rhythm for at least 30 minutes. Patients who have not converted by the time 3 DC shocks have been delivered or who revert to AF/AFL during the 30 minutes following the shocks will be considered treatment failures. Spontaneous conversion after randomization but prior to study interventions will be considered a treatment success.

SECONDARY OUTCOMES:
Outcomes during ED Visit | 1 day
  Being in normal sinus rhythm at the time of ED disposition

OTHER OUTCOMES:
ED disposition | 1 day
  ED disposition - admission or discharge;
Length of stay in ED | 1 day
  Length of stay in ED in minutes from time of arrival to time of discharge or admission
Time to conversion to sinus rhythm | 1 day
  Time to conversion to sinus rhythm in minutes from time of randomization; a 60 minute adjustment will be made for those randomized to placebo infusion.
Adverse Events | 1 day
  Adverse events:
  i) conduction problems: development of new bundle branch block or QT lengthening >25% from baseline; ii) dysrhythmias: bradycardia (heart rate < 50 bpm), ventricular tachyarrhythmias (torsade de pointes, sustained ventricular tachycardia > 30 seconds, or ventricular fibrillation), or cardiac arrest; iii) hypotension: systolic BP < 90 mm-Hg; iv) respiratory events: hypoxia (O2 saturation < 90%), aspiration, or airway manoeuvres (e.g., jaw positioning, oral airway, BVM ventilation, intubation).
Physician Comments | 1 month
  Physician comments on the protocol gathered as narrative by research staff.

CONTACTS AND LOCATIONS:
Overall Officials: Ian G Stiell, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (10):
- Canada (10):
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital Du Sacre-Coeur, Montreal, Quebec
  - Hopital de L'Enfant-Jesus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stiell IG, Sivilotti MLA, Taljaard M, Birnie D, Vadeboncoeur A, Hohl CM, McRae AD, Morris J, Mercier E, Macle L, Brison RJ, Thiruganasambandamoorthy V, Rowe BH, Borgundvaag B, Clement CM, Brinkhurst J, Brown E, Nemnom MJ, Wells GA, Perry JJ. A randomized, controlled comparison of electrical versus pharmacological cardioversion for emergency department patients with acute atrial flutter. CJEM. 2021 May;23(3):314-324. doi: 10.1007/s43678-020-00067-7. Epub 2021 Jan 18. PMID 33959925
- [Derived] Stiell IG, Sivilotti MLA, Taljaard M, Birnie D, Vadeboncoeur A, Hohl CM, McRae AD, Rowe BH, Brison RJ, Thiruganasambandamoorthy V, Macle L, Borgundvaag B, Morris J, Mercier E, Clement CM, Brinkhurst J, Sheehan C, Brown E, Nemnom MJ, Wells GA, Perry JJ. Electrical versus pharmacological cardioversion for emergency department patients with acute atrial fibrillation (RAFF2): a partial factorial randomised trial. Lancet. 2020 Feb 1;395(10221):339-349. doi: 10.1016/S0140-6736(19)32994-0. PMID 32007169